CLINICAL TRIAL: NCT01429311
Title: Investigation of Reduced Interferon Responses in Peripheral Blood Mononuclear Cells of Participants With Atopic Dermatitis and a History of Eczema Herpeticum (ADRN-01)
Brief Title: Interferon Responses in Eczema Herpeticum
Acronym: ADRN-01
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Atopic Dermatitis Research Network (Other)
Responsible Party: Sponsor
Other Study IDs: DAIT ADRN-01; NIAID Funding Mechanism (Other Grant/Funding Number: HHSN272201000020C and HHSN272201000017C)
Record Dates: First submitted 2011-07-19; First posted 2011-09-07 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Atopic Dermatitis; Eczema Herpeticum; Herpes Simplex Infections; Eczema Vaccinatum
Keywords: Atopic Dermatitis; Eczema herpeticum; Interferon gamma; IFNγ
MeSH Terms: conditions — Dermatitis, Atopic; Kaposi Varicelliform Eruption; Herpes Simplex

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples, RNA, serum, protein and cells will be retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- ADEH+: Subjects classified as Atopic Dermatitis (AD) and history of previous Eczema Herpeticum (EH) as defined by the ADRN Standard Diagnostic Criteria
- ADEH-: Subjects classified as AD without a history of EH as defined by the ADRN Standard Diagnostic Criteria
- Non-atopic Controls: Subjects classified as "Non-Atopic controls" as defined by the ADRN Standard Diagnostic Criteria

SUMMARY:
Atopic dermatitis (AD) is a chronic skin disorder characterized by recurrent viral skin infections. A small subset of patients with AD suffer from disseminated viral infections, e.g., eczema herpeticum (ADEH+), after herpes simplex infection (HSV) or eczema vaccinatum (EV) after smallpox vaccination. Interferon gamma (IFNγ) plays a critical role in the innate and acquired immune responses by activating macrophages, enhancing natural killer cell activation, and promoting T cell differentiation, as well as regulating B cell isotype switching to immunoglobulin (Ig) G2a. Recent studies have demonstrated that IFNγ generation was significantly decreased after stimulation with HSV ex vivo. The purpose of this study is to determine if deficient IFNγ induction leads to susceptibility to HSV infection in ADEH+ patients.

DETAILED DESCRIPTION:
The investigators hypothesize that defective IFNγ responses in peripheral blood mononuclear cells (PBMCs) from ADEH+ patients results from aberrant pattern recognition receptors (PRR) signaling in antigen-presenting cells (APCs) resulting in low level production of IL-12, an essential cytokine for IFNγ generation. This study will compare results from 40 ADEH+, 40 ADEH-, and 40 non-atopic participants.

Study procedures will typically be completed in one visit; however, participants may be asked to return for additional unscheduled visit(s) occurring as frequently as every 3 months for the duration of the study to provide an additional blood sample for further characterization of immune mechanisms leading to reduced IFNγ responses in ADEH+.

ELIGIBILITY:
Participant Inclusion Criteria:

Participants who meet all of the following criteria are eligible for enrollment:

* have a history of AD with or without a history of Eczema Herpeticum (EH) as diagnosed using the Atopic Dermatitis Research Network (ADRN) Standard Diagnostic Criteria OR

  --are non-atopic as diagnosed using the ADRN Standard Diagnostic Criteria
* are willing to sign the informed consent form or whose parent or legal guardian is willing to sign the informed consent form (age appropriate) prior to initiation of any study procedure
* are willing to sign the assent form, if age appropriate.

Participant Exclusion Criteria:

Participants who meet any of the following criteria are not eligible for enrollment:

* have a history of any systemic illness (e.g., immunodeficiency disorders such as human immunodeficiency virus [HIV] or lupus erythematosus) other than the condition being studied
* have an active systemic malignancy, excluding uncomplicated non-melanoma skin cancer
* have any skin disease other than AD that might compromise the stratum corneum barrier (e.g., bullous disease, psoriasis, cutaneous T cell lymphoma [also called Mycosis Fungoides or Sezary syndrome], dermatitis herpetiformis, Hailey-Hailey, or Darier's disease)
* have a first degree relative already enrolled in the study
* are determined not to be eligible in the opinion of the Investigator.

Participants who meet any of the following criteria are not eligible for enrollment but may be reassessed:

* have active eczema herpeticum at the Enrollment Visit
* have taken systemic immunosuppressive drugs including cyclosporine or oral steroids within 30 days of the Enrollment Visit
* have a fever ≥ 38.5 degrees Centigrade (ºC) (101.3 ºF) at the Enrollment Visit.

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 40 ADEH+, 40 ADEH-, and 40 non-atopic controls ages 6 to 65 years. Initially, 20 ADEH- and 20 non-atopic control participants will be gender- and age-matched (plus or minus 10 years) to 20 ADEH+ participants. Afterwards, additional participants will be enrolled such that the gender ratio and the age distribution of the ADEH+ participants will be similar to that of the ADEH- and non-atopic control participants
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2011-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Expression of IFNγ and Interleukin-12 (IL-12), in response to stimulation with Herpes Simplex Virus 1 (HSV-1), Vaccinia Virus (VV), and Pattern Recognition Receptors (PRR) agonists | Day 1
  Protein and messenger ribonucleic acid (mRNA) levels of IFNγ, and the IFN-γ promoting cytokine, IL-12, produced by Cluster of Differentiation 14 (CD14+) monocytes in response to stimulation with HSV-1, VV, and various PRR agonists

SECONDARY OUTCOMES:
Cell surface expression of Major Histocompatibility complex (MHC) class I and class II and co-stimulatory molecules on CD14+ cells in response to IFNγ and Interferon-alpha (IFNα) stimulation | Day 1
Production of IL-18 and IFNα protein and mRNA by CD14+ cells following stimulation with HSV-1, VV, or PRR agonists | Day 1
Production of IFNγ protein by Cluster of Differentiation 8 (CD8+) T cells in response to stimulation with recombinant human cytokines including but not limited to IL-12, IL-18, and IFNα | Day 1
Protein expression of IFNγ receptor and IFNα/β receptor on CD14+ cells | Day 1
Immunodominant HSV-1 peptide repertoires | Day 1
  Analysis of immunodominant HSV-1 peptide repertoires with related Human Leukocyte Antigen (HLA) in ADEH+, ADEH-, and non-atopic participants
High-throughput gene expression profiling to analyze ribonucleic acid (RNA) from HSV-1 stimulated and sham stimulated CD14+ monocytes | Day 1
  Global transcriptional response of CD14+ monocytes to stimulation with HSV-1 as evaluated by GeneChip Profiling
Production of protein and RNA of IFN family members and any related pro- or anti-inflammatory cytokines/chemokines in response to stimulation of PBMCs or purified monocytes | Day 1
  IFN family members include IFNα, Interferon beta (IFNβ), and IFNγ. Related pro- or anti-inflammatory cytokines/chemokines include, but are not limited to IL-29 and IL-10
Expression of MHC and co-stimulatory molecules on CD14+ cells in response to stimulation with HSV-1, VV, or PRR agonists | Day 1
Viral titer of VV as determined by plaque assay following incubation of virus with PBMCs | Day 1
Gene expression profiles and gene variant profiles of PBMCs stimulated with HSV-1 as assayed by RNA-seq | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Donald Leung, PhD, M.D, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

REFERENCES:
- [Result] Gao L, Bin L, Rafaels NM, Huang L, Potee J, Ruczinski I, Beaty TH, Paller AS, Schneider LC, Gallo R, Hanifin JM, Beck LA, Geha RS, Mathias RA, Barnes KC, Leung DYM. Targeted deep sequencing identifies rare loss-of-function variants in IFNGR1 for risk of atopic dermatitis complicated by eczema herpeticum. J Allergy Clin Immunol. 2015 Dec;136(6):1591-1600. doi: 10.1016/j.jaci.2015.06.047. Epub 2015 Sep 3. PMID 26343451
- [Result] Bin L, Edwards MG, Heiser R, Streib JE, Richers B, Hall CF, Leung DY. Identification of novel gene signatures in patients with atopic dermatitis complicated by eczema herpeticum. J Allergy Clin Immunol. 2014 Oct;134(4):848-55. doi: 10.1016/j.jaci.2014.07.018. Epub 2014 Aug 23. PMID 25159465
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait